CLINICAL TRIAL: NCT02829177
Title: A Double-blind, Randomized, Placebo Controlled Trial of Allopurinol in Patients With Type 1 Diabetes and Microalbuminuria
Brief Title: Microalbuminuria and Allopurinol in Type 1 Diabetes
Acronym: MIKAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peter Rossing (Other)
Responsible Party: Sponsor-Investigator, Peter Rossing, Senior Principal Investigator, Professor, Chief Physician, DMSc, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 3004
Record Dates: First submitted 2015-03-27; First posted 2016-07-12 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Type 1 Diabetes; Diabetic Nephropathy
Keywords: Type 1 diabetes; Diabetic nephropathy; Albuminuria; Allopurinol
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Nephropathies; Albuminuria | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allopurinol (Active Comparator): 400 mg once daily, tablet treatment
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator): Identical tablet treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allopurinol
  Arms: Allopurinol
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective is to determine if lowering serum uric acid by means of allopurinol in the course of kidney disease may be effective in preventing or improving albuminuria and renal function in Type 1 Diabetic patients. The study is a double blinded, randomised, placebo-controlled cross-over clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Albuminuria (≥30 mg/g)
* Uric Acid ≥ 0,265 mmol/l
* GFR (glomerular filtration rate) > 40 ml/min/1.73m2

Exclusion Criteria:

* History of gout or xanthinuria or other indications for uric acid lowering therapy such as cancer chemotherapy.
* Recurrent renal calculi.
* Current use of azathioprine, 6-mercaptopurine, didanosine, tamoxifen, amoxicillin/ampicillin, or other drugs interacting with allopurinol.
* Known allergy to xanthine-oxidase inhibitors.
* Renal transplant.
* Non-diabetic kidney disease.
* Home, 24h og clinical BP>180 or Diastolic BP >130 mmHg at screening.
* Cancer treatment within two years before screening.
* History of hepatitis B or C.
* History of acquired immune deficiency syndrome or human immunodeficiency virus (HIV) infection.
* History of alcohol or drug abuse.
* Breastfeeding or pregnancy or unwillingness to be on contraception throughout the trial.
* Poor mental function or any other reason to expect patient difficulty in complying with the requirements of the study.
* Serious pre-existing medical problems other than diabetes, e.g. congestive heart failure, pulmonary insufficiency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2016-08-10 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Improved Albuminuria | 60 days
  Improvement of albuminuria will be evaluated by the collection of 24h urin collection with the measure of 24h albumine excretion rate and the measurements will be compared for the two treatment arm for each participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No